CLINICAL TRIAL: NCT01619813
Title: A Randomized Phase II Study of Reolysin in Combination With Docetaxel and Prednisone or Docetaxel and Prednisone Alone in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Reolysin Combined With Docetaxel and Prednisone or Docetaxel and Prednisone Alone in Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Oncolytics Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I209
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; reolysin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docetaxel, Reolysin and Prednisone (Active Comparator)
  Interventions: Drug: Docetaxel, Reolysin and Prednisone
- Docetaxel and Prednisone (Active Comparator)
  Interventions: Drug: Docetaxel and Prednisone

INTERVENTIONS:
Drug: Docetaxel, Reolysin and Prednisone — Docetaxel 75 mg/m2 will be delivered as a 1-hour infusion q 3 weekly beginning on day 1, cycle 1. Reolysin will be delivered as a 1-hour infusion days 1-5. On day 1 of each cycle, when both agents are given, the docetaxel will be given first. Prednisone 5 mg BID will be given beginning day 1. Each cycle is 3 weeks in length.
  Arms: Docetaxel, Reolysin and Prednisone
Drug: Docetaxel and Prednisone — Docetaxel 75 mg/m2 will be delivered as a 1-hour infusion q 3 weekly. Prednisone 5mg BID will be given beginning Day 1. Each cycle is 3 weeks in length.
  Arms: Docetaxel and Prednisone

SUMMARY:
The purpose of this study is to find out if giving Reolysin in combination with docetaxel and prednisone can offer better results than standard therapy with docetaxel and prednisone.

DETAILED DESCRIPTION:
Researchers doing this study also want to evaluate the side effects of Reolysin when given together with docetaxel and prednisone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological diagnosis of adenocarcinoma of the prostate.
* All patients must have a formalin fixed paraffin embedded tissue block (from their primary or metastatic tumour) available for translational studies.
* Presence of clinically and/or radiologically documented disease (measurable or non-measurable). All radiology studies must be performed within 28 days prior to randomization (within 35 days if negative). Patients with elevated PSA only are not eligible.
* Androgen ablation must include either medical or surgical castration. If the patient is receiving medical androgen ablation, a castrate level of testosterone (< 1.7 nmol/L) must be present.
* Patients must have metastatic or locally recurrent disease, for which no curative therapy exists and for which systemic therapy is indicated due to progression following castration.

Progression is defined as one or both of the following:

PSA Progression:

A rising PSA, while receiving androgen ablative therapy, with 2 subsequent rises over a reference value (not necessarily consecutively), measured a minimum of one week apart. The PSA that confirms progression must have a value of ≥2 ng/ml and must be performed no longer than 7 days prior to trial randomization. Patients who have had prolonged responses to combined androgen blockade should be evaluated for a withdrawal response prior to confirming eligibility OR

Radiological Progression:

defined as the development of new metastatic lesions or progression in target disease (RECIST 1.1) with a stable or rising PSA.

* The PSA must be ≥ 5 ng/ml at the time of study entry.
* ECOG performance of 0, 1 or 2.
* Age ≥ 18 years of age.
* Patients must have a life expectancy of ≥ 12 weeks.
* Previous Therapy

Surgery:

Previous major surgery is permitted provided that it has been at least 14 days prior to patient randomization and that wound healing has occurred.

Chemotherapy:

Patients may NOT have received any prior cytotoxic chemotherapy for recurrent/metastatic castration resistant prostate cancer. Prior docetaxel treatment is not permitted unless it was provided on an adjuvant therapy protocol more than 12 months prior to study enrollment.

Hormonal Therapy:

Prior hormone therapy is required. Patients must be castrate resistant and have discontinued anti-androgens for at least 4 weeks prior to study entry (at least 6 weeks for bicalutamide). Therapy with LHRH agonist must continue for those prostate cancer patients already receiving this treatment at the time of enrollment. If the patient has discontinued the LHRH agonist, this must be restarted (if not surgically castrated) and the castrate level of testosterone must be present. Prior therapy with CYP17 inhibitors (e.g. abiraterone, ketoconazole) or novel anti-androgens (e.g. MDV3100) is permitted.

Radiation:

Prior external beam radiation is permitted provided a minimum of 4 weeks has elapsed between the last dose and enrollment to the trial. Exceptions may be made for low dose, non-myelosuppressive radiotherapy after consultation with NCIC CTG. Prior strontium is not permitted.

* Laboratory Requirements (must be done within 7 days prior to randomization)

Hematology:

Granulocytes (AGC) ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L

Biochemistry:

Serum creatinine ≤ 1.5 x ULN Total bilirubin ≤ 1.0 x ULN (unless elevated secondary to conditions such as Gilbert's disease) ALT and AST ≤ 1.5 x ULN Proteinuria <2g/24hrs (screen using spot testing; if ≥ grade 2 repeat with mid-stream urine - if still ≥ grade 2 then urine collection for 24 hours to confirm <2g/24hrs)

* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.

Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients) are not to be recruited into the study. Patients competent but physically unable to sign the consent form may have the document signed by their nearest relative or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.

* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 2 hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves that the patients registered on this trial will be available for complete documentation of the treatment, adverse events, response assessment and follow-up.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient randomization.

Exclusion Criteria:

* Patients with a history of other malignancies, except for adequately treated non-melanoma skin cancer or solid tumours curatively treated with no evidence of disease for ≥ 3 years.(Please call NCIC CTG if any questions about the interpretation of this criterion).
* Patients who are on immunosuppressive therapy or have known HIV infection or active hepatitis B or C.
* Patients with active or uncontrolled infections, or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
* Patients are not eligible if they have a known hypersensitivity to the study drug(s) or their components.
* Patients with history of central nervous system metastases or untreated spinal cord compression.
* Patients who have had prior treatment with docetaxel for advanced/metastatic disease.
* Men who are not sterile unless they use an adequate method of birth control.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-12-14 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2016-05-20 (Actual)

PRIMARY OUTCOMES:
Disease Progression | 12 weeks
  Efficacy will be based on the lack of disease progression measured at 12 weeks.

SECONDARY OUTCOMES:
Effect of Docetaxel and Reolysin on circulating tumour cells | 12 weeks
  Effect of docetaxel and Reolysin on the circulating tumour cell (CTC) favourable status (< 5 CTC per 7.5mL). Effect will be measured after 6 and 12 weeks of treatment.
PSA change rate | 24 months
Objective Response | 24 months
  Objective response rate (in patients with measurable disease at baseline)
Overall Survival | 24 months
Determine patient tolerability and toxicity of Reolysin and Docetaxel in combination | 24 months
  Determine the effect of Reolysin and Docetaxel in combination in patients.
Prognostic/Predictive molecular response | 24 months
  Explore potential molecular factors which might be prognostic/predictive of response (tumour, CTCs, serial blood samples).

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Eigl, Study Chair — BCCA Vancouver
Locations (11):
- Canada (11):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Abbotsford Centre, Abbotsford, British Columbia
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eigl BJ, Chi K, Tu D, Hotte SJ, Winquist E, Booth CM, Canil C, Potvin K, Gregg R, North S, Zulfiqar M, Ellard S, Ruether JD, Le L, Kakumanu AS, Salim M, Allan AL, Feilotter H, Theis A, Seymour L. A randomized phase II study of pelareorep and docetaxel or docetaxel alone in men with metastatic castration resistant prostate cancer: CCTG study IND 209. Oncotarget. 2018 Jan 17;9(8):8155-8164. doi: 10.18632/oncotarget.24263. eCollection 2018 Jan 30. PMID 29487723